CLINICAL TRIAL: NCT07135245
Title: Improved Treatment and Monitoring of Alzheimer's Disease - a Randomized Controlled Clinical Trial
Brief Title: Improved Treatment and Monitoring of Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rune Skovgaard Rasmussen (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Rune Skovgaard Rasmussen, MSc, PhD, associate professor of General Pathology, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 523376
Record Dates: First submitted 2025-08-04; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease (AD)
Keywords: Alzheimer Disease; Semaglutide; Cognition; Dental care; retinal hyper-reflective foci
MeSH Terms: conditions — Alzheimer Disease | interventions — semaglutide; candesartan; Calcium

STUDY DESIGN:
Intervention Model Description: 180 participants with mild cognitive impairments are randomized into 3 groups of 60 participants each and treated for 1.5 years (78 weeks):
  1. An intervention group treated with semaglutide (Rybelsus®) 3 mg daily for 4 weeks followed by 7 mg daily for 4 weeks, hereafter 14 mg daily and placebo.
  2. An intervention group will be treated with semaglutide (Rybelsus®) 3 mg daily for 4 weeks, followed by 7 mg daily for 4 weeks, and subsequently 14 mg daily. The intervention will also include candesartan up to 32 mg daily, a multivitamin-mineral tablet containing vitamin D and calcium, increased oral hygiene and a tooth lozenge (CariGuard®).
  3. A control group treated with placebo and no further intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment with medications will be double blinded and oral hygiene treatment will be single blinded, as it is impossible to blind patients to increased oral hygiene. The evaluators of a patient do not know the patient's treatment group, or if it is a baseline evaluation or a final evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention - semaglutide only (Experimental): An intervention group treated with semaglutide (Rybelsus®) 3 mg daily for 4 weeks followed by 7 mg daily for 4 weeks, hereafter 14 mg daily and placebo.
  Interventions: Drug: Semaglutide (Rybelsus®)
- Control (Placebo Comparator): A control group treated with placebo and no further intervention.
  Interventions: Other: Placebo
- Intervention - combination (Experimental): An intervention group will be treated with semaglutide (Rybelsus®) 3 mg daily for 4 weeks, followed by 7 mg daily for 4 weeks, and subsequently 14 mg daily. The intervention will also include candesartan up to 32 mg daily, a multivitamin-mineral tablet containing vitamin D and calcium, increased oral hygiene and a tooth lozenge (CariGuard®).
  Interventions: Drug: Semaglutide (Rybelsus®) combined with other interventions

INTERVENTIONS:
Drug: Semaglutide (Rybelsus®) combined with other interventions — The full intervention includes treatment with semaglutide (Rybelsus®) 3 mg daily for 4 weeks, followed by 7 mg daily for 4 weeks, and subsequently 14 mg daily. The intervention will also include candesartan up to 32 mg daily, a multivitamin-mineral tablet containing vitamin D and calcium, increased oral hygiene and a tooth lozenge (CariGuard®)
  Other Names: Candesartan, multivitamin-mineral tablets containing vitamin D and calcium, increased oral hygiene and a tooth lozenge (CariGuard®); Combination group
  Arms: Intervention - combination
Other: Placebo — A control group treated with placebo and no further intervention
  Arms: Control
Drug: Semaglutide (Rybelsus®) — An intervention group treated with semaglutide (Rybelsus®) 3 mg daily for 4 weeks followed by 7 mg daily for 4 weeks, hereafter 14 mg daily and placebo
  Arms: Intervention - semaglutide only

SUMMARY:
In the world's high-income countries, Alzheimer's disease and other dementia diseases are currently the second most common cause of death. This is a recent change, as strokes in the form of blood clots or bleedings in the brain previously were the second most common cause of death.

In Denmark 90,000 live with dementia and life expectancy after dementia diagnosis is 5 to 8 years. Of these, 50,000 have Alzheimer's disease. By 2040 due to a steep increase of the elderly population, the number of people with dementia in Denmark is expected to profoundly increase to 120,000-146,000. This is a concerning forecast which calls for action for several reasons. First and foremost, for the sake of the many thousands of persons who will experience dementia. Every three hours, a Dane dies of dementia. There is currently no cure for Alzheimer's disease and there is a need for the development of an effective therapy. The use of cholinesterase inhibitors, such as donepezil, galantamine and rivastigmine, and the NMDA receptor antagonist memantine, may relieve symptoms, but cannot stop disease progression.

Glucagon-like peptide-1 (GLP-1) receptor agonists (RAs) are among the promising therapies for repurposing as a treatment for Alzheimer's disease. Dementia rate was significantly lower both in type 2 diabetic patients randomized to GLP-1 RAs versus placebo (hazard ratio: 0.47) and in a nationwide Danish registry-based cohort (HR: 0.89) with yearly increased exposure to GLP-1 RAs in a publication on pooled data from three randomized double-blind placebo-controlled trials (15,820 patients) and the cohort (120,054 patients). It is not known whether treatment with GLP-1 RAs may reduce the incidence of dementia in patients without diabetes. There are ongoing studies of whether the GLP-1 RA semaglutide (Rybelsus®), which has a 94% similarity to the naturally occurring human GLP-1 hormone, has a positive effect on early Alzheimer's disease, namely the EVOKE and EVOKE Plus clinical trials.

In this present placebo-controlled clinical trial, the effect of semaglutide (Rybelsus®) on cognitive impairment in Alzheimer's disease will be investigated. The primary hypothesis is that treatment with semaglutide (Rybelsus®) in combination with other treatments will reduce the progression of the cognitive impairment compared to the control group. In comparison with the EVOKE trials focusing on semaglutide as monotherapy, this present trial will investigate the effect of semaglutide both alone and combined with other treatments.

The secondary hypothesis is that patients with mild cognitive impairment and Alzheimer's disease have a more frequent incidence of gingivitis and periodontitis, especially with the bacterium Porphyromonas gingivalis producing its toxins in the oral cavity. Recent research has indicated that this bacteria from the mouth and gingiva through the bloodstream can spread to the brain and be a trigger for Alzheimer's disease. Lactobacillus rhamnosus (LGG) has demonstrated to decrease the level of Porphyromonas gingivalis in plaque along with reduction in gingivitis.

Further hypotheses tested in this trial

* Administration of candesartan to patients with biomarker-confirmed initial-stage Alzheimer's disease will decrease levels of amyloid markers, improve cognitive function, and enhance brain connectivity.
* Daily multivitamin-mineral, including vitamin D and calcium supplementation, will improve global cognition, episodic memory, and executive functions in older adults.
* Alzheimer's disease is associated with certain abnormalities of vision and of the structure of the visual system, both of which can precede the development of symptoms of cognitive decline. Hard drusen are yellow deposits under the retina typically made up of lipids and proteins, which may predict retinal pathology, were more commonly found in the temporal region of Alzheimer's disease retinas compared to retinas of normal older patients. Retinal nerve fiber layer thickness will be measured, retinal drusen, retinal hyper-reflective foci, and foveal avascular zone area in patients with treated Alzheimer's disease compared to controls.
* Gait analysis will be performed and may be particularly sensitive to early symptoms of dementia development.
* • Biomarkers (p-beta-amyloid, p-tau217 and p-tau181) in cerebrospinal fluid (CSF) will be measured to support suspected Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Decreased cognitive abilities corresponding to 16-25 points in the Mini Mental State Examination (MMSE)
* The cognitive impairment must be supported by the presence of specific levels in cerebrospinal fluid (CSF) of β-Amyloid1-42 (≤1030 pg/ml) and Tau (total and phosphorylated, respectively over 300 pg/ml and 27 pg/ml)
* MRI scan of the brain with coronal sections showing substance loss (atrophy) of the medial part of the temporal lobe compatible with Alzheimer's disease
* PET scan of the brain (18F-FDG PET) with decreased regional glucose metabolism in the temporal and parietal regions and PiB (PiB-PET scan) with amyloid plaques in the brain compatible with Alzheimer's disease

Exclusion Criteria:

* Patients with active cancer, and in chemo- or radiation therapy
* Severe cardiovascular disease.
* Hepatic insufficiency with ASAT> 2 x upper limit of normal or renal insufficiency with serum creatinine > 200 micromol/l
* Severe epilepsy with frequent tonic-clonic (grand mal) seizures
* Insulin treatment (type 1 diabetes mellitus) and diabetic ketoacidosis
* Severe chronic disease (e.g., cirrhosis, AIDS, chronic kidney failure)
* Severe mental illness e.g., schizophrenia, or physical disabilities leading to inability to participate in intervention or tests, or to provide informed consent
* Evidence for other primary causes of neurodegeneration or dementia, e.g., significant cerebrovascular disease (whose primary cause of dementia was vascular in origin), Lewy Body disease, Parkinson's disease, Fronto-temporal dementia
* Significant ongoing psychiatric or substance abuse problems.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
The Montreal Cognitive Assessment | At inclusion, and 52 and 78 weeks.
  The Montreal Cognitive Assessment is a cognitive screening instrument which provides an estimate of the level of intellectual functioning. Scores are from 0 to 30, where a score of 26 or higher is considered normal. Montreal Cognitive Assessment is moreover sensitive to mild cognitive problems as well as dementia. Studies have shown that Montreal Cognitive Assessment is more sensitive than Mini Mental State Examination to detecting mild cognitive changes and is as effective in identifying the incidence of Alzheimer's disease.

SECONDARY OUTCOMES:
Measurement of β-Amyloid1-42 | Performed at inclusion, and 6, 12, and 18 months.
  Measurement in CSF of β-Amyloid1-42 using the Elecsys System Cobas® provided by Roche Diagnostics, Denmark, where more pronounced changes in markers for positive identification of Alzheimer's disease in the control group will be expected. Measurements of beta-amyloid, vitamin D and Herpes Simplex Virus (HSV-1) will be carried out by the medical investigator.
Measurement of Tau | At inclusion, and 6, 12, and 18 months
  Measurement in CSF of Tau (total and phosphorylated) using the Elecsys System Cobas® provided by Roche Diagnostics, Denmark, where more pronounced changes in markers for positive identification of Alzheimer's disease in the control group will be expected. CSF levels of phosphorylated p-tau217 and p-tau181 are measured at inclusion and thereafter every 6 months.
MRI scan of the brain | At inclusion, and 52 and 78 weeks.
  Registration of substance loss (atrophy) of the medial part of the temporal lobe demonstrated in coronal sections, compatible with Alzheimer's disease, will be performed, and patients will be monitored for other kinds of brain pathologies. We will use resting state fMRI data to analyze trends of functional connectivity alterations in the patients.
PET scan of the brain | At inclusion, and 52 and 78 weeks.
  PET scans will be performed using (18F-FDG PET) to identify any decreased regional glucose metabolism in the temporal and parietal regions and PiB (PiB-PET scan) with amyloid plaques in the brain compatible with Alzheimer's disease.
Clinical Dementia Rating scale - Sum of Boxes | At inclusion, and 52 and 78 weeks.
  Clinical Dementia Rating scale - Sum of Boxes (CDR-SB) scores reliably discriminated between mild cognitive impairment (MCI) and very early Alzheimer disease.The CDR-SB provides a more quantitative measure than the single "Global CDR Score." It is considered more sensitive to early cognitive changes and is useful for tracking changes over time, especially in clinical trials. General guidelines for interpreting the CDR-SB score are as follows:
  0: Normal 0.5 - 4.0: Questionable cognitive impairment to very mild dementia 4.5 - 9.0: Suggests mild dementia 9.5 - 15.5: Suggests moderate dementia 16.0 - 18.0: Suggests severe dementia
Symbol Digit Modalities Test | At inclusion, and 52 and 78 weeks
  Danish norms exists. Participants are given a key showing a set of geometric symbols and their corresponding digits (e.g., a "]" symbol corresponds to the number "4"). They then have a grid of symbols and must quickly write or say the correct digit for each symbol. The test is timed, with a standard duration of 90 seconds. The raw score is simply the total number of correct substitutions made within that 90-second interval. Incorrect or omitted responses do not count. Higher scores are better.
Quality of Life - Alzheimer's Disease (QoL-AD). | At inclusion, and 52 and 78 weeks
  The Quality of Life-Alzheimer's Disease (QoL-AD) scale is a widely used tool for assessing the subjective well-being of individuals with Alzheimer's and other forms of dementia. It is scored in a straightforward manner, but its key feature is that it can be completed by both participants and caregivers (proxy), which allows for a more comprehensive view of their quality of life.
  The QoL-AD consists of 13 items covering various life domains, such as physical health, energy, mood, living situation, memory, family, friends, and the ability to do things for fun. Each of the 13 items is rated on a 4-point scale:
  1. = Poor
  2. = Fair
  3. = Good
  4. = Excellent
  The total score is the sum of the ratings for all 13 items. The minimum possible score is 13 (1 point for each of the 13 items), and the maximum is 52 (4 points for each item). A higher score indicates a better quality of life.
Patient Global Impression of Change (PGI-C). | At inclusion, and 52 and 78 weeks
  The Patient Global Impression of Change (PGI-C) is a single-item, patient-reported outcome measure used to evaluate a patient's overall perception of how their condition has changed since the start of a treatment or study. Scoring is based on a simple, usually 7-point, Likert scale.
  The PGI-C is a self-administered questionnaire that asks the patient to rate the change in their condition. The scale ranges from "very much worse" to "very much improved," with "no change" as the midpoint.
  Instead of a total score like other scales, the PGI-C result is a single number corresponding to the patient's selected response. The interpretation is often dichotomous, meaning it's used to classify patients into "improved" or "not improved." The PGI-C is considered a "gold standard" for assessing a subjective experience of change because it directly asks them what participants think. This is useful in clinical trials to complement objective measures and provide participant-centered perspectives.
European Quality of Life-5 Dimensions Questionnaire (EuroQol-5D™, EQ-5D) | At inclusion, and 52 and 78 weeks
  The EuroQol-5 Dimensions (EQ-5D) is a widely used, standardized instrument for measuring health-related quality of life. It is scored in two main parts, which are often used independently or together: the descriptive system and the EQ Visual Analogue Scale (EQ VAS).
  The responses to the five dimensions are combined into a 5-digit code or "health profile." For example, a response of "no problems," "slight problems," "moderate problems," "severe problems," and "extreme problems" would be represented by the health profile 12345 on the EQ-5D-5L. A score of 11111 represents perfect health. A descriptive health profile (e.g., 11123), which can be converted into a single index value (utility score) using a country-specific value set.
  The EQ Visual Analogue Scale (EQ VAS) is a separate, single-item component of the EQ-5D, where participants are asked to rate their overall health "today" on a vertical scale from 0 to 100. The score is simply the number the respondent marks on the scale..
The Major Depression Inventory (MDI) | At inclusion, and 52 and 78 weeks.
  The Major Depression Inventory (MDI) is a self-report questionnaire used to assess depressive symptoms and the severity of depression. As a severity scale, MDI provides a total score that indicates the degree of depressive symptoms. Total Score: The scores from all 10 items are summed up. The theoretical range of the total score is from 0 (no depression) to 50 (maximum depression).
The Rey-Osterrieth Complex Figure Test | At inclusion, and 52 and 78 weeks.
  The Rey-Osterrieth Complex Figure (ROCF) test is a neuropsychological assessment used to evaluate visuospatial abilities, memory, and executive functions. Participants copy an advanced visual figure (without later recall). Rey-Osterrieth Complex Figure is scored by a trained clinician who systematically evaluates the accuracy and placement of 18 specific components, with a maximum possible score of 36, higher scores are best. This process provides a quantitative measure of visuospatial and memory skills and a qualitative understanding of the individual's cognitive strategy. Danish norms exist. The test is sensitive to Alzheimer's disease.
The 12-item Neuropsychiatric Inventory (NPI-12) | At inclusion, and 52 and 78 weeks.
  The 12-item Neuropsychiatric Inventory (NPI-12) is scored based on a structured interview with a caregiver who knows the patient well. Only the Caregiver Distress Scale will be used. For each of 12 symptom domain where a behavior is present, the caregiver is asked to rate how distressing the behavior is for them personally.
  Distress Rating: This is rated on a scale from 0 to 5:
  0: Not distressing at all
  1. Minimal
  2. Mild
  3. Moderate
  4. Severe
  5. Extreme or very severe
  The Total Caregiver Distress Score range from 0 (best) to 60 (worst). This score helps researchers understand the impact of the patient's behaviors on their caregivers.

IPD SHARING:
Plan to Share IPD: Undecided